CLINICAL TRIAL: NCT06244446
Title: Efficacy and Safety of SBRT Combined With Atezolizumab Plus Bevacizumab vs Atezolizumab Plus Bevacizumab in Treating Unresectable Advance Hepatocellular Carcinoma (SAB - A Prospective Observational Study).
Brief Title: Efficacy and Safety of SBRT Combined With Atezolizumab Plus Bevacizumab vs Atezolizumab Plus Bevacizumab in Treating Unresectable Advance Hepatocellular Carcinoma.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-HCC-07
Record Dates: First submitted 2024-01-10; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, stool, urine & saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBRT+Atezolizumab+Bevacizumab
  Interventions: Other: No intervention
- Atezolizumab+Bevacizumab
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention. It is an observational study

SUMMARY:
SBRT, atezolizumab, and bevacizumab have different mechanisms of action and can potentially have synergistic effects when combined. SBRT delivers targeted radiation to the tumor, while atezolizumab enhances the immune response, and bevacizumab inhibits angiogenesis. The combination of SBRT with atezolizumab and bevacizumab will result in improved tumor response rates as compared to atezolizumab and bevacizumab alone in patients with advance unresectable hepatocellular carcinoma (HCC). Up until now, no study has been done that has compared SBRT with atezolizumab, and bevacizumab in unresectable advance hepatocellular carcinoma. With this study, investigator aim to study to compare the efficacy and safety of SBRT combined with atezolizumab and bevacizumab versus atezolizumab and bevacizumab alone in the treatment of unresectable advance hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Hypothesis: The combination of SBRT with atezolizumab and bevacizumab will result in improved tumor response rates as compared to atezolizumab and bevacizumab alone in patients with advance unresectable hepatocellular carcinoma (HCC).

AIM:- The aim of this study is to compare the efficacy and safety of SBRT combined with atezolizumab and bevacizumab versus atezolizumab and bevacizumab alone in the treatment of unresectable advance hepatocellular carcinoma (HCC).

Study design:

* A prospective observational study.
* Single Centre.
* Open label.
* The study will be conducted in Department of Hepatology, ILBS. Study period: 1 years after ethical approval.

Sample size:

* Assuming that objective response rate with immunotherapy is 30%, further adding SBRT along with immunotherapy is increased by 50% that is objective response rate by adding SBRT is 80% .
* With ⍺-5 and power 80%, investigator need to enroll 36 cases and further adding 10% dropout rate investigator need to enroll 40 cases i.e. 20 in each group.

Monitoring and assessment: All the parameters of the objective and also noted any adverse effects.

Intervention: Nil

STATISTICAL ANALYSIS:

The continuous data will be represented as mean +/- SD or median (IQR). The categorical data will be represented as median (IQR).The comparison of continuous data will be done by using either Student's t test or Mann -Whitney test as appropriate. The Kaplan Meier and Cox regression will be used for survival analysis. Besides this an appropriate analysis will be done at the time of data analysis. P value < 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age; 18-70 years.
2. Unresectable advance HCC with PVTT
3. At least one measurable (measurable according to Response Evaluation Criteria In Solid Tumors (mRECIST V.1.1)), untreated lesions.
4. Patients with hepatitis B virus (HBV) infection: HBV-DNA <500 IU/mL obtained within 28 days before the start of study treatment and received anti-HBV treatment for at least 28 days before entering the study.
5. Patients with hepatitis C virus (HCV) infection: HCV-DNA <500 IU/mL obtained within 28 days before the start of study treatment and received anti-HCV treatment for at least 28 days before entering the study.
6. Maximum diameter of tumor ≤ 15cm
7. Maximum number of tumor nodules ≤5
8. Liver function: Child-Pugh class A, B7; normal liver volume is more than 800cm3.
9. Karnofsky performance status ≥ 80%
10. The expected survival of the patient is more than 6 months.
11. Agree to accept post-procedure follow-up required by the design of this study.
12. The following conditions are met:

    i. Platelet≥60×109/L; White blood cell≥3.0×109/L; Hemoglobin≥85 g/L; Serum creatinine≤1.4 × upper limit;. PT-INR ≤1.7

Exclusion Criteria:

1. Patients with untreated or incompletely treated esophageal and/or gastric varices with associated bleeding or at high risk of bleeding.
2. Coinfection with HBV and hepatitis C virus (HCV).
3. Symptomatic, untreated or progressively progressive central nervous system (CNS) metastases.
4. The patient cannot receive follow-up or is participating in other clinical trials.
5. Subjects deemed unsuitable for inclusion in this study by the investigator.
6. Current or past autoimmune disease or immunodeficiency.
7. History of leptomeningitis.
8. Idiopathic pulmonary fibrosis, organising pneumonia or evidence of active pneumonia on chest.
9. Known active tuberculosis.
10. Severe infection within 4 weeks prior to initiation of study treatment
11. A potential subject who meets any of the following criteria will be excluded from participation in this study:

    i) Previous radiotherapy to the liver ii) Known current pregnancy iii) Loss of fat planes of tumor with organ at risk like the esophagus, stomach, duodenum, small bowel on CT or on MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC with PVTT (BCLC -C)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR), which is defined as the proportion of patients with complete response (CR) and partial response (PR) at 6 months . CR or PR is assessed in accordance with mRECIST. | 6 months

SECONDARY OUTCOMES:
Overall survival | 3 months.
Overall survival | 6 months.
Overall survival | 12 months.
Disease control rate (DCR) at 3 months, defined as the percentage of subjects with the best response as CR, PR or stable disease (SD). | 3 months.
Disease control rate (DCR) at 6 months, defined as the percentage of subjects with the best response as CR, PR or stable disease (SD). | 6 months.
Disease control rate (DCR) at12 months, defined as the percentage of subjects with the best response as CR, PR or stable disease (SD). | 12 months.
Progression-free survival (PFS) | 3 months.
Progression-free survival (PFS) | 6 months.
Progression-free survival (PFS) | 12 months.
Adverse events | 3 months.
Adverse events | 6 months.
Adverse events | 12 months.
Number of Participants with biomarkers change ( AFP , PIVKA II) in both groups. | 3 months.
Number of Participants with biomarkers change ( AFP , PIVKA II) in both groups. | 6 months.
Number of Participants with biomarkers change ( AFP , PIVKA II) in both groups. | 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No